CLINICAL TRIAL: NCT06007235
Title: A Randomized, Double-Blind, Placebo-Controlled, Crossover, Pilot Stage Clinical Trial Evaluating CACIPLIQ20 in Wound Healing in Subjects With Epidermolysis Bullosa
Brief Title: CACIPLIQ20 in Wound Healing in Subjects With Epidermolysis Bullosa
Acronym: MATHBULL
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Organ, Tissue, Regeneration, Repair and Replacement (Industry)
Collaborators: Euraxi Pharma (Industry); ARANZ Medical (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Quadruple | Purpose: Supportive Care
Other Study IDs: 2022-A01774-39
Record Dates: First submitted 2023-08-07; First posted 2023-08-23 (Actual); Last update posted 2024-02-13 (Actual); Status verified 2024-02

CONDITIONS: Epidermolysis Bullosa Dystrophica; Epidermolysis Bullosa, Junctional
MeSH Terms: conditions — Epidermolysis Bullosa Dystrophica; Epidermolysis Bullosa, Junctional

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: Blinding codes on treatments
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- A: CACIPLIQ20 before placebo (Other): Arm A will receive at first CACIPLIQ20 (experimental product) for 1 month, followed by 1-month washout, then 1 month of saline (placebo comparator).
  Interventions: Device: CACIPLIQ20; Drug: Placebo
- B: placebo before CACIPLIQ20 (Other): Arm B will receive at first saline (placebo comparator) for 1 month, followed by 1-month washout, then 1 month of CACIPLIQ20 (experimental product).
  Interventions: Device: CACIPLIQ20; Drug: Placebo

INTERVENTIONS:
Device: CACIPLIQ20 — CACIPLIQ20 contains RGTA heparan sulphate mimetics
Drug: Placebo — Saline solution in identical spray bottles

SUMMARY:
Epidermolysis bullosa (EB) is a group of inherited disorders characterized by fragility of the skin and mucous membranes within the basement membrane zone. It is characterized by moderate to excessive fragility of epithelial tissues with prototypic blistering or erosions following minimal trauma (mechanobullous dermatoses). The chronic pain associated with EB, the hardship placed on caregivers, and the high risk for complications places a considerable psychosocial burden on both patients and their families. Despite considerable research to advance the understanding of EB pathophysiology, no treatments have been approved by regulatory authorities to date.

Heparan sulfates are key elements of the Extra Cellular Matrix scaffold which act both as linkers, bridging structural matrix proteins such as collagens, laminin and as storage and protector sites to communication peptides, playing a pivotal role in the regulation of cell proliferation, migration and differentiation that are all required for tissue regeneration and repair. CACIPLIQ20 is a bioengineered structural analogue of heparan sulfate glycosaminoglycans. Numerous experimental studies have provided strong evidence that CACIPLIQ20 promotes tissue regeneration by reconstructing the cellular microenvironment following tissue injury. CACIPLIQ20 is currently a class III CE marked medical device (NSAI-0050 CE MARK ECDECNL-A4 (6) and EC Annex II of the directive. NL-A4 (7)) with the following indications: Chronic ulcers showing no tendency to heal after 6 months of standard care, or still unhealed after 12 months:

* Pressure ulcers.
* Peripheral arterial disease (such as Stage IV Leriche & Fontaine) ulcers.
* Diabetic ulcers (including amputation).

Preliminary results from several published and unpublished case reports (Al Malak and Barritault, 2012; Bodemer, unpublished observations) suggest that CACIPLIQ20 is safe and can improve wound healing and reduce pain in patients with epidermolysis bullosa.

The goal of the MATHBULL study is to confirm preliminary observations in a placebo-controlled double-blind pilot study. The results of this pilot study will help to design a pivotal study.

DETAILED DESCRIPTION:
The patients are outpatients at inclusion and may be already followed by the investigators, and they have not yet been treated with CACIPLIQ20 for at least one month.

These patients will be randomly allocated (1:1 ratio) to Arm A and B. Every patient will have two treatment periods. Arm A will receive at first CACIPLIQ20 for 1 month, followed by 1-month washout then 1-month Placebo, and the reverse sequence (Placebo followed by CACIPLIQ20) in Arm B. The sponsor, investigator and patient will remain blinded to the treatment Arm in which a patient will be randomized until the end of the study and database lock.

Two baselines will be defined before the two treatment periods, Baseline 1 at inclusion/before treatment period 1, and Baseline 2 at the end of washout/before treatment period 2.

For each patient, all active wounds will be treated by CACIPLIQ20 or Placebo, which will be added to the best standard of care decided by the participating physicians. Treatments will be provided in indistinguishable spray bottles, labelled with treatment numbers using a randomization list provided by an independent statistician. CACIPLIQ20 or Placebo will be applied every 3 to 4 days for 30 days. Patients will be followed every month according to investigators' standard practices. At least five visits will be programmed during the study, including Inclusion Visit, End of Treatment Period 1 Visit at Month 1, End of Washout Visit at Month 2, End of Treatment Period 2 Visit at Month 3, End of Study Visit at Month 4. In addition to these visits, two phone calls will be organized 15 days after the start of each treatment period to identify potential adverse events.

At each visit, the investigator will take pictures of treated wounds with an imaging device (Silhouette®), in order to assess the total lesioned skin surface.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of Dystrophic or Junctional EB.
* 3 years ≤ age ≤ 18 years
* At least one active wound at inclusion
* Informed consent form signed by the patient's legal representative; if the patient is minor but capable of providing consent, additional signed consent from the patient.
* Patient and caregiver must be willing to comply with all protocol requirements.

Exclusion Criteria:

* Use of any investigational drug within the last 30 days before enrolment.
* Current or former malignancy.
* Pregnancy or breastfeeding during the study.
* Females of childbearing potential who are not abstinent and not practicing a medically acceptable method of contraception.
* Use of CACIPLIQ20 within the last 30 days before enrolment.
* Patients intolerant to one of the study device components or to heparinoids.

Ages: 3 Years to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 16 (Estimated)
Dates: Start 2024-01-29 (Actual); Primary Completion 2024-09 (Estimated); Study Completion 2024-09 (Estimated)

PRIMARY OUTCOMES:
Change in total lesioned skin surface | After 1 month of treatment
  Change in total lesioned skin surface from baseline* to the end of the CACIPLIQ20 vs Placebo treatment periods
  * Baseline 1 at inclusion/before treatment period 1, and Baseline 2 at the end of washout/before treatment period 2 Change in total lesioned skin surface at the end of each treatment period will be assessed blindly regarding treatment allocation, using the SilhouetteConnect™ software in reference to "Baseline 1" and "Baseline 2".

SECONDARY OUTCOMES:
The rate of device related serious adverse events | Up to 4 months
The rate of device related adverse events | Up to 4 months
The rate of procedure related adverse events | Up to 4 months
The rate of procedure related serious adverse events | Up to 4 months
The rate of all adverse events (AEs). | Up to 4 months
The rate of all serious adverse events (SAE) | Up to 4 months
Proportion of wounds achieving complete closure at the end of the CACIPLIQ20 versus Placebo treatment periods | After 1 month of treatment
  This parameter will be assessed with the ARANZ Silhouette® system by comparing wounds areas before and after each treatment period.
Mean CGI at the end of the CACIPLIQ20 versus Placebo treatment periods | After 1 month of treatment
  The CGI (clinical assessment) will be rated on the following sevenpoint scale:
  1. = Very much improved-nearly all better; good level of functioning; minimal symptoms; represents a very substantial change
  2. = Much improved-notably better with significant reduction of symptoms; increase in the level of functioning but some symptoms remain
  3. = Minimally improved-slightly better with little or no clinically meaningful reduction of symptoms. Represents very little change in basic clinical status, level of care, or functional capacity
  4. = No change-symptoms remain essentially unchanged
  5. = Minimally worse-slightly worse but may not be clinically meaningful; may represent very little change in basic clinical status or functional capacity
  6. = Much worse-clinically significant increase in symptoms and diminished functioning
  7. = Very much worse-severe exacerbation of symptoms and loss of functioning
Mean SGI at the end of the CACIPLIQ20 versus Placebo treatment periods | After 1 month of treatment
  The SGI (subject/family assessment) will be rated on the following sevenpoint scale:
  1. = Very much improved-nearly all better; good level of functioning; minimal symptoms; represents a very substantial change
  2. = Much improved-notably better with significant reduction of symptoms; increase in the level of functioning but some symptoms remain
  3. = Minimally improved-slightly better with little or no clinically meaningful reduction of symptoms. Represents very little change in basic clinical status, level of care, or functional capacity
  4. = No change-symptoms remain essentially unchanged
  5. = Minimally worse-slightly worse but may not be clinically meaningful; may represent very little change in basic clinical status or functional capacity
  6. = Much worse-clinically significant increase in symptoms and diminished functioning
  7. = Very much worse-severe exacerbation of symptoms and loss of functioning
Change in pain assessed from baseline to the end of the CACIPLIQ20 versus Placebo treatment periods (for patients from 3 to 4 years of age) | After 1 month of treatment
  Change in pain will be assessed at the end of the one-month treatment period 1 and 2 compared to baseline 1 and baseline 2, respectively, using the "FLACC scale" for patients from 3 to 4 years of age.
  FLACC: Face Legs Activity Cry Consolability. Score range for the FLACC scale is between 0-10 where higher score represents more pain.
Change in pain assessed from baseline to the end of the CACIPLIQ20 versus Placebo treatment periods (for patients 4 years of age and older) | After 1 month of treatment
  Change in pain will be assessed at the end of the one-month treatment period 1 and 2 compared to baseline 1 and baseline 2, respectively, using the "Wong Faces Pain Scale" for patients 4 years of age and older.
  The Wong Faces Pain Scale rates pain on a 0-10 scale, where higher score represents more pain.
Change in itching assessed from baseline to the end of the CACIPLIQ20 versus Placebo treatment periods | After 1 month of treatment
  Change in itching will be assessed at the end of one-month treatment period 1 and 2 with eference to baseline 1 and baseline 2, respectively. Itching will be measured using the "Itch Man Pruritus Assessment Tool". In patients from 3 to 6 years of age, assessments will be performed by caretakers whereas patients who are 6 years of age and older will self-report their itching using the "Itch Man Pruritus Assessment Tool".
  Itching assessments based on the following scores: 0=Comfortable, no itch; 1=itches a little, does not interfere with activity; 2=itches more, sometimes interferes with activity; 3=itches a lot, difficult to be still, concentrate; 4=itches most terribly, impossible to sit still or concentrate.

CONTACTS AND LOCATIONS:
Overall Officials: Christine Bodemer, MD, PhD, Principal Investigator — Hopital Necker - enfants malades
Locations (1):
- Hopital Necker - enfants malades, Paris, France

IPD SHARING:
Plan to Share IPD: Undecided